CLINICAL TRIAL: NCT00427258
Title: An Open-Label, Single-Dose Study of the Mass Balance and Metabolic Disposition of Orally Administered [14C]MOA-728 in Healthy Men
Brief Title: Study Evaluating MOA-728 Administered in Healthy Men
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3200A3-1106
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: healthy subjects

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
Absorption, distribution, metabolism, and excretion (ADME) study with 14C in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 50 years inclusive at screening.
* Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight ≥50 kg. BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's height, in meters, at screening: BMI = weight (kg)/[height (m)]2
* Healthy as determined by the investigator on the basis of screening evaluations.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01

PRIMARY OUTCOMES:
Distribution of drug using radioactive study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.